CLINICAL TRIAL: NCT04580654
Title: A 2-Part, Phase 1, Single Center, Open-label, Single Ascending Dose Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Subcutaneous and Intravenous CSL312 in Healthy Adult Japanese and Caucasian Subjects
Brief Title: A Study to Assess the Pharmacokinetics and Safety of CSL312 in Healthy Japanese and Caucasian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CSL312_1003
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CSL312 (Cohort 1a, low dose) (Experimental): Factor XIIa antagonist monoclonal antibody administered subcutaneously
  Interventions: Biological: CSL312
- CSL312 (Cohort 1b, low dose) (Experimental): Factor XIIa antagonist monoclonal antibody administered subcutaneously
  Interventions: Biological: CSL312
- CSL312 (Cohort 2, high dose) (Experimental): Factor XIIa antagonist monoclonal antibody administered subcutaneously
  Interventions: Biological: CSL312
- CSL312 (Cohort 3, low dose) (Experimental): Factor XIIa antagonist monoclonal antibody administered intravenously
  Interventions: Biological: CSL312
- CSL312 (Cohort 4, high dose) (Experimental): Factor XIIa antagonist monoclonal antibody administered intravenously
  Interventions: Biological: CSL312

INTERVENTIONS:
Biological: CSL312 — Fully human immunoglobulin G4/lambda recombinant monoclonal antibody against Factor XIIa
  Other Names: Factor XIIa antagonist monoclonal antibody; garadacimab

SUMMARY:
This will be a 2- part, phase 1, open-label, single center, single ascending dose study to investigate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of subcutaneous (SC) and intravenous (IV) administration of CSL312 in healthy adult Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian and Japanese male or female subjects 18 to 55 years old (inclusive) that meet the following criteria at Screening:

  * Japanese subjects defined as being born in Japan, having not lived outside of Japan for more than 10 years, and having both parents and four grandparents who are of Japanese ancestry.
  * Caucasian subjects, defined as having both parents and four grandparents descended from and of the peoples of Europe, the Middle East, or North Africa, who are body weight-matched (± 15%) 1:1 with Japanese subjects.
* Body weight in the range of ≥ 50 kg and ≤ 100 kg
* Body mass index of ≥ 18 kg/m2 and ≤ 30 kg/m2

Exclusion Criteria:

* Positive serology test for human immunodeficiency virus (HIV)-1 / 2 antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis C virus (HCV) antibody.
* Received any live viral or bacterial vaccinations within 8 weeks of Screening or is expected to receive any live virus or bacterial vaccinations during the study.
* Evidence of current active infection.
* Known malignancy or a history of malignancy in the past 5 years .
* Blood pressure or pulse rate measurements outside the normal range for the subject's age.
* Female subject of childbearing potential or fertile male subject either not using or not willing to use an acceptable method of contraception
* Pregnant, breastfeeding, or not willing to cease breastfeeding.
* Donation or loss of more than 500 mL of blood within 3 months, or donated plasma within 7 days
* History of clinically significant arterial or venous thrombosis, bleeding disorder, or any abnormal coagulation test result

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Area under the curve (AUC) from time 0 extrapolated to infinity (AUC0-inf) of CSL312 after subcutaneous dosing | Up to 85 days postdose

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-last) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Half-life (t1/2) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Apparent clearance (CL/F) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Apparent volume of distribution (Vz/F) of CSL312 after subcutaneous dosing | Up to 85 days postdose
Cmax of CSL312 after intravenous dosing | Up to 85 days postdose
Tmax of CSL312 after intravenous dosing | Up to 85 days postdose
AUC0-last of CSL312 after intravenous dosing | Up to 85 days postdose
AUC0-inf of CSL312 after intravenous dosing | Up to 85 days postdose
t1/2 of CSL312 after intravenous dosing | Up to 85 days postdose
Clearance (CL) of CSL312 after intravenous dosing | Up to 85 days postdose
Volume of distribution (Vd) of CSL312 after intravenous dosing | Up to 85 days postdose
Mean FXIIa-mediated kallikrein activity | Up to 85 days postdose
Number of subjects experiencing adverse events (AEs) | Up to 85 days postdose
Percentage of subjects experiencing AEs | Up to 85 days postdose
Number of subjects experiencing serious adverse events (SAEs) | Up to 85 days postdose
Percentage of subjects experiencing SAEs | Up to 85 days postdose
Number of subjects experiencing adverse events of special interest (AESIs) | Up to 85 days postdose
Percentage of subjects experiencing AESIs | Up to 85 days postdose
Number of subjects experiencing Anti-CSL312 antibodies | Up to 85 days postdose
Percentage of subjects experiencing Anti-CSL312 antibodies | Up to 85 days postdose
Number of subjects with injection / infusion site reaction by severity | Up to 48 hours after start of infusion or injection
Percentage of subjects with injection / infusion site reaction by severity | Up to 48 hours after start of infusion or injection

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.